CLINICAL TRIAL: NCT07351643
Title: Assessment of the Effects of SGLT2 Inhibitors on Pericoronary Fat in Non-diabetic ACS Patients Without Heart Failure Using CCTA
Brief Title: CCTA Evaluation of SGLT2i-related Pericoronary Fat Changes in Non-diabetic ACS Patients Without HF
Acronym: DAPA-PCAT
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shenyang Northern Hospital (Other)
Responsible Party: Principal Investigator, Han Yaling, Prof., Shenyang Northern Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYNH-Y2025503; Y(2025)503 (Other: Northern Theater Command General Hospital Ethics Committee)
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: ACS (Acute Coronary Syndrome); SGLT2 Inhibitors
Keywords: Fat attenuation index; SGLT2 inhibitors; Pericoronary adipose tissue; Residual inflammatory risk; Coronary CT angiography
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: Eligible participants will undergo CCTA at 1 month after PCI. Those meeting all criteria will then be randomized 1:1 to the dapagliflozin group or standard care group using a dynamic block randomization method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dapagliflozin group (Experimental): Participants receive dapagliflozin 10 mg orally once daily in addition to guideline-directed medical therapy for 6 months.
  Interventions: Drug: Dapagliflozin
- Non-dapagliflozin group (No Intervention): Participants receive guideline-directed medical therapy alone without any SGLT2 inhibitor for 6 months.

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg/d for 6 months
  Arms: Dapagliflozin group

SUMMARY:
The goal of this clinical trial is to learn if dapagliflozin, a sodium-glucose cotransporter 2 inhibitor (SGLT2i), can reduce coronary artery inflammation in people with acute coronary syndrome (ACS) who do not have diabetes or heart failure.

Coronary inflammation will be measured using the fat attenuation index (FAI), a marker derived from coronary CT angiography (CCTA) that quantifies inflammation in the fat tissue surrounding heart arteries.

The main questions it aims to answer are:

* Does dapagliflozin lower coronary artery inflammation as measured by FAI?
* Does dapagliflozin slow the progression of coronary plaques?

Researchers will compare participants who take dapagliflozin 10 mg daily plus standard therapy to those who receive standard therapy alone for 6 months.

Participants will:

* Undergo percutaneous coronary intervention (PCI) for ACS
* Have a baseline CCTA scan at 1 month after PCI, at which point they will be randomly assigned to receive dapagliflozin or standard care alone
* Have a follow-up CCTA scan at 6 months after randomization
* Have blood tests at the time of PCI, at randomization, and at 6 months after randomization
* Receive follow-up phone calls at 3 and 6 months after randomization

DETAILED DESCRIPTION:
SCIENTIFIC BACKGROUND

Residual inflammatory risk (RIR) has emerged as a major driver of adverse cardiovascular outcomes in patients with acute coronary syndrome (ACS), even after guideline-directed medical therapy and successful revascularization. Recent pooled analyses of the PROMINENT, REDUCE-IT, and STRENGTH trials demonstrated that high-sensitivity C-reactive protein (hsCRP), a marker of RIR, predicts future cardiovascular events more strongly than LDL-cholesterol in statin-treated patients.

Pericoronary adipose tissue (PCAT) fat attenuation index (FAI), measured by coronary CT angiography (CCTA), has been validated as a novel imaging biomarker that directly quantifies coronary artery inflammation. When coronary inflammation occurs, PCAT undergoes characteristic morphological changes with decreased lipid content and increased water-to-fat ratio, resulting in higher CT attenuation values (shifting from approximately -190 Hounsfield Units toward -30 HU). The CRISP-CT study validated this imaging biomarker and demonstrated its prognostic value for cardiac mortality independent of conventional cardiovascular risk factors.

SGLT2 inhibitors have established cardiovascular benefits in patients with diabetes or heart failure. Beyond glucose-lowering and diuretic effects, anti-inflammatory mechanisms may contribute to these benefits, including suppression of inflammatory cytokines such as interleukin-6 and monocyte chemoattractant protein-1, reduction of oxidative stress, and improvement of endothelial function. Clinical studies have shown that SGLT2 inhibitors reduce epicardial adipose tissue volume and may stabilize coronary plaques in diabetic patients. The EMPA-TROPISM study provided evidence that empagliflozin reduces epicardial adipose tissue volume even in non-diabetic patients with heart failure, suggesting glucose-independent mechanisms.

KNOWLEDGE GAP

The EMPACT-MI and DAPA-MI trials recently evaluated SGLT2 inhibitors in patients with acute myocardial infarction without diabetes or heart failure, with primary endpoints focused on clinical outcomes. Neither trial specifically assessed coronary inflammation using validated imaging biomarkers. Whether SGLT2 inhibitors exert measurable anti-inflammatory effects at the coronary arterial level in this population remains unknown.

STUDY RATIONALE

This study addresses this knowledge gap by employing CCTA-derived pericoronary fat attenuation index as a direct measure of coronary inflammation. The study population specifically excludes patients with diabetes and heart failure to isolate the potential anti-inflammatory effects of dapagliflozin from its established benefits in these conditions. Assessment of non-culprit vessels in patients with multivessel disease allows longitudinal evaluation of atherosclerotic changes without interference from prior intervention.

STUDY TIMELINE

Participants undergo PCI for ACS at enrollment. At 1 month post-PCI, eligible participants undergo baseline CCTA and are then randomized to receive either dapagliflozin plus standard therapy or standard therapy alone. This timing allows for stabilization of the acute coronary event before baseline imaging assessment. Follow-up CCTA is performed at 6 months post-randomization to evaluate changes in FAI and plaque characteristics.

CLINICAL SIGNIFICANCE

Current anti-inflammatory therapies for secondary prevention of coronary artery disease have significant limitations, including high cost and limited accessibility for monoclonal antibodies such as canakinumab, and gastrointestinal side effects with poor tolerability for low-dose colchicine. If this study demonstrates that SGLT2 inhibitors reduce coronary inflammation in non-diabetic patients without heart failure, it would expand therapeutic options for addressing residual inflammatory risk and potentially benefit a broader patient population beyond those with diabetes or heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Diagnosis of acute coronary syndrome (including ST-elevation myocardial infarction, non-ST-elevation myocardial infarction, or unstable angina)
3. Undergoing percutaneous coronary intervention (PCI)
4. Presence of multivessel coronary artery disease with at least one non-culprit vessel not undergoing revascularization (for CCTA follow-up assessment)
5. Willing and able to provide written informed consent

Exclusion Criteria:

1. Prior or current diagnosis of diabetes mellitus
2. Prior or current diagnosis of chronic heart failure
3. Treatment with any SGLT2 inhibitor within 4 weeks prior to enrollment
4. Severe hepatic impairment
5. History of recurrent urogenital infections
6. Known allergy or intolerance to SGLT2 inhibitors
7. Pregnancy or breastfeeding
8. Systolic blood pressure <90 mmHg and/or diastolic blood pressure <60 mmHg
9. Severe chronic kidney disease (eGFR <30 mL/min/1.73 m²)
10. Current participation in another interventional clinical trial
11. Any other condition that, in the opinion of the investigator, would make the participant unsuitable for enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2026-02-25 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in FAI from baseline to 6 months in patients assessed by CCTA | From randomization to 6 months post-randomization
  Change in FAI of major coronary arteries (left main [LM], right coronary artery [RCA], left anterior descending [LAD], and left circumflex [LCX]) from baseline to 6 months, expressed in Hounsfield Units (HU), assessed at the patient level.

SECONDARY OUTCOMES:
Change in total plaque volume | From randomization to 6 months post-randomization
  Absolute change in total coronary plaque volume (mm³)
Change in calcified plaque volume | From baseline (at randomization) to 6 months post-randomization
  Absolute change in calcified plaque volume (mm³)
Change in fibrous plaque volume | From baseline (at randomization) to 6 months post-randomization
  Absolute change in fibrous plaque volume (mm³)
Change in fibrofatty plaque volume | From baseline (at randomization) to 6 months post-randomization
  Absolute change in fibrofatty plaque volume (mm³)
Change in low-attenuation plaque volume | From baseline (at randomization) to 6 months post-randomization
  Absolute change in low-attenuation plaque volume (mm³)
Change in coronary stenosis | From baseline (at randomization) to 6 months post-randomization
  Absolute change in degree of coronary artery stenosis (%)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Northern Theater Command, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No